CLINICAL TRIAL: NCT06153069
Title: Clinical Efficacy of a Short-course Regimen for Asymptomatic Tuberculosis in China
Brief Title: Asymptomatic TB With Innovative Modified Short-course Regimens
Acronym: SWIFT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2023-715
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Tuberculosis
Keywords: subclinical tuberculosis; shorter treatment
MeSH Terms: conditions — Tuberculosis | interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Four-month regimen (Experimental): The four-month regimen consists of a 17-week course of standard daily first-line anti-tuberculosis therapy, administered as either fixed-dose combinations or separate bulk drugs, in accordance with the recommendations of Technical Guidelines for Tuberculosis Prevention and Control in China. The treatment comprises an intensive phase of 8 weeks with Isoniazid (H) , Rifampicin (R), Pyrazinamide (Z) and Ethambutol (E), followed by continuation phase of 9 weeks with HR. If the sputum culture remains positive at week 8, or if the radiological examination at the end of treatment still shows unclosed cavities, the continuation phase treatment will be extended by an additional 8 weeks.
  Interventions: Drug: Four-month regimen
- Standardized Regimen (Active Comparator): The standardized regimen consists of a 26-week course of standard daily first-line anti-tuberculosis therapy, administered as either fixed-dose combinations or separate bulk drugs, in accordance with the recommendations of Technical Guidelines for Tuberculosis Prevention and Control in China. The treatment comprises an intensive phase of 8 weeks with Isoniazid (H) , Rifampicin (R), Pyrazinamide (Z) and Ethambutol (E), followed by continuation phase of 18 weeks with HR.
  Interventions: Drug: Standard regimen
- Three-month regimen (Experimental): Three-month regimen consists of two periods of 13-21 weeks. During the intensive phase (8 weeks), rifapentine 900 mg daily; moxifloxacin 400 mg daily; isoniazid 300 mg daily; pyrazinamide <50.0kg 1000mg daily, 50.0-70.9kg 1500 mg daily, ≥71kg 2000mg daily. During the continuation phase (5 or 13 weeks based on the culture resultes and radiological manifestations), rifapentine 900 mg daily; moxifloxacin 400 mg daily; isoniazid 300 mg daily; All treatment is taken orally. For rifapentine administration, the daily dosage may be reduced to 600mg if intolerance occurs.
  Interventions: Drug: Three-month regimen

INTERVENTIONS:
Drug: Four-month regimen — The four-month regimen consists of a 17-week course of standard daily first-line anti-tuberculosis therapy, administered as either fixed-dose combinations or separate bulk drugs, in accordance with the recommendations of Technical Guidelines for Tuberculosis Prevention and Control in China. The treatment comprises an intensive phase of 8 weeks with Isoniazid (H) , Rifampicin (R), Pyrazinamide (Z) and Ethambutol (E), followed by continuation phase of 9 weeks with HR. If the sputum culture remains positive at week 8, or if the radiological examination at the end of treatment still shows unclosed cavities, the continuation phase treatment will be extended by an additional 8 weeks.
  Arms: Four-month regimen
Drug: Three-month regimen — Three-month regimen consists of two periods of 13-21 weeks. During the intensive phase (8 weeks), rifapentine 900 mg daily; moxifloxacin 400 mg daily; isoniazid 300 mg daily; pyrazinamide <50.0kg 1000mg daily, 50.0-70.9kg 1500 mg daily, ≥71kg 2000mg daily. During the continuation phase (5 or 13 weeks based on the culture resultes and radiological manifestations), rifapentine 900 mg daily; moxifloxacin 400 mg daily; isoniazid 300 mg daily; All treatment is taken orally. For rifapentine administration, the daily dosage may be reduced to 600mg if intolerance occurs.
  Arms: Three-month regimen
Drug: Standard regimen — The standardized regimen consists of a 26-week course of standard daily first-line anti-tuberculosis therapy, administered as either fixed-dose combinations or separate bulk drugs, in accordance with the recommendations of Technical Guidelines for Tuberculosis Prevention and Control in China. The treatment comprises an intensive phase of 8 weeks with Isoniazid (H) , Rifampicin (R), Pyrazinamide (Z) and Ethambutol (E), followed by continuation phase of 18 weeks with HR.
  Arms: Standardized Regimen

SUMMARY:
This study is a randomized controlled trial among asymptomatic tuberculosis individuals aiming to assess whether the standard treatment duration can be shortened to 17 weeks without increasing the types or doses of anti-tuberculosis medications or 13 weeks with the high-dose rifapentine and moxifloxacin.

DETAILED DESCRIPTION:
This study is a prospective, open-label, multicenter randomized controlled trial. The randomization process will use centralized stratified block randomization to minimize bias across province of participating sites.

Asymptomatic tuberculosis individuals included in the study will be randomly assigned in a 1:1:1 ratio to three groups: Standard Regimen Group, Four-month Regimen Group or Three-month Regimen Group. The standard regimen consists of rifampicin (R), isoniazid (H), pyrazinamide (Z), and ethambutol (E) for 8 weeks, followed by rifampicin and isoniazid for an additional 18 weeks. The four-month regimen group follows the same regimen as the standard regimen group for the initial 8 weeks, followed by a continuation phase of daily rifampin (R) and isoniazid (H) for 9 weeks. The three-month regimen consists of high-dose rifapentine (P), isoniazid (H), pyrazinamide (Z), and moxifloxacin (M) for 8 weeks, followed high-dose Rifapentine (P), isoniazid (H), and moxifloxacin (M) for 5 weeks. For individuals in the four-month and the three-month regimen group, the treatment response will be evaluated at the end of the treatment phase. If the sputum culture remains positive at week 8, or if the radiological examination at the end of treatment still shows unclosed cavities, the continuation phase treatment will be extended by an additional 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 14 to 80 years;
* 2. Male or female;
* 3. Willing to provide signed informed consent, or parental consent and participant assent;
* 4. Individuals with respiratory tract specimen (including sputum/bronchoalveolar lavage fluid/lung tissue) positive for acid-fast bacilli smear/culture/molecular amplification for M. tuberculosis;
* 5. No unexplained TB-suggestive symptoms in the three months prior to screening, including cough lasting more than two weeks, night sweats, fever or weight loss;
* 6. If non-menopausal woman, agree to use or have used effective contraception during treatment.

Exclusion Criteria:

* 1. Combined extrapulmonary tuberculosis;
* 2. Induviduals with extensive lesion (lesion involvement exceeding 50% or the aggregate diameter of all cavities exceeding 6 cm) ;
* 3. Individuals will be excluded from enrollment if, at the time of enrollment, their M. tuberculosis isolate is already known to be resistant to any one or more of the following: rifampin, isoniazid, pyrazinamide, ethambutol, or fluoroquinolones;
* 4. Individuals with impaired liver function (alanine transaminase [ALT] or total bilirubin [TBIL] more than 2.5 times the upper limit of normal) or combined with liver cirrhosis;
* 5. Hemoglobin is less than 70g/L, or platelet is less than 50*10^9/L;
* 6. Estimated Glomerular Filtration Rate (eGFR) is less than 30 mL/min/1.73m2;
* 7. Known allergic or intolerant to any of the study drugs;
* 8. Pregnant or breast-feeding;
* 9. Prior anti-TB treatment for more than one week in the past six months;
* 10.Known history of epilepsy, uncontrolled diabetes;
* 11.For HIV-positive subjects, T-lymphocyte (CD4 cell) counts less than 100 cells/mm3;
* 12. Unable to tolerant oral treatment.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 426 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Favorable outcome rate in mITT pupulation | At 78 weeks post-randomization
  To compare the proportion of participants in mITT population achieving favorable outcome at 78 weeks post-randomization.

SECONDARY OUTCOMES:
Favorable outcome rate in assessable and PP population | At 78 weeks post-randomization
  To compare the proportion of participants in assessable population and PP population achieving favorable outcomes at 78 weeks post-randomization.
Relapse rate post-treatment | At 104 weeks post-randomization
  To compare the proportion of relapse rate post-treatment.
The proportion of participants with sputum culture conversion | At 8 weeks post-randomization
  The proportion of participants with sputum culture conversion at 8 weeks post-randomization
The proportion of grade 3 or greater adverse events | From treatment initiation until two weeks after the last dose
  To evaluate the proportion of participants who experience grade 3 or greater adverse events.
Acquired drug resistance | Post-treatment follow-up phase
  The proportion of participants acquiring drug resistance during follow-up.
Acceptability to regimens | At the end of treatment
  The total score of acceptability in mITT population and PP population at the end of treatment.
The overall index score of quality of life | At the end of treatment and at 78 weeks post-randomization
  The overall index score of quality of life in mITT population and PP population at the end of treatment and at 78 weeks post-randomization.
Community transmission risk | From treatment initiation
  The community transmission risk in mITT and PP population.
Serious adverse events | From informed consent through final follow-up
  Proportion of serious adverse events from the date of informed consent until completion of the final follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, Dr., Principal Investigator — Huashan Hospital of Fudan University，Shanghai，China
Locations (5):
- China (5):
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Liupanshui City Third People's Hospital, Liupanshui, Guizhou
  - Nayong County People's Hospital, Nayong, Guizhou
  - Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The First People's Hospital of Linping District, Hangzhou, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR